CLINICAL TRIAL: NCT03335176
Title: Feasibility and Benefit of a Telerehabilitation Program in Human Immunodeficiency Virus-infected Patients
Brief Title: Feasibility of Telerehabilitation in HIV-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Caty, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telerehabilitation HIV
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance and Resistance Training Exercise (Experimental)
  Interventions: Behavioral: Endurance ad Resistance Training Exercise
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Endurance ad Resistance Training Exercise — Patients received a 6-week tele-supervised rehabilitation with 3 exercise sessions per week
  Arms: Endurance and Resistance Training Exercise

SUMMARY:
The aim of this study is to assess the feasibility and the effects of a 6-week telerehabilitation on the three domains of the International Classification of Functioning, Disability and Health in HIV-infected patients under highly active antiretroviral therapy (HAART).

HIV-infected patients were randomized either into an Endurance and Resistance Training Exercise (ERTE) group or a control (CON) group. Telerehabilitation was realized in a public fitness center, with online guidance and weekly telephone advice, 3 times per week for 6 weeks. Feasibility was determined by recruitment rate, retention rate and adverse events. Secondary outcomes were impact on body composition, inflammation and coagulation (C-reactive protein, D-dimer), physical fitness and quality of life (WHOQOL-HIV).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* under HAART treatment
* native French speaker

Exclusion Criteria:

* AIDS diagnosis
* physical and/or psychiatric impairments that seriously impaired physical activity
* pregnant
* Unstable (defined by any modification of health outcomes during the last 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At study completion (after 6 weeks)
  Number of eligible participants who enrolled in the program out of the number were recruited
Retention rate | At study completion (after 6 weeks)
  Percentage of patients lost to follow-up
Adverse events | At study completion (after 6 weeks)
  Percentage of patients who experienced one or more adverse events

SECONDARY OUTCOMES:
Weight | Assessments at baseline and at 6 weeks
  Weight (kg) is measured by using a bioelectrical impedance analysis
Lean body mass | Assessments at baseline and at 6 weeks
  Lean body mass (kg) is measured by using a bioelectrical impedance analysis
Fat body mass | Assessments at baseline and at 6 weeks
  Lean body mass (kg) is measured by using a bioelectrical impedance analysis
C-reactive protein | Assessments at baseline and at 12 weeks
  C-reactive protein is measured by a blood test
D-dimer | Assessments at baseline and at 12 weeks
  D-dimer is measured by a blood test
CD4+ T cell counts | Assessments at baseline and at 12 weeks
  CD4+ T cell counts is measured by a blood test
Viral load | Assessments at baseline and at 12 weeks
  Viral load is measured by a blood test
Functional exercise capacity | Assessments at baseline and at 6 weeks
  Functional exercise capacity is measured by a 6-minute walk test
Flexibility | Assessments at baseline and at 6 weeks
  Flexibility is measured by Toe touch test and sit and reach test
Lower body muscular strength | Assessments at baseline and at 6 weeks
  Lower body muscular strength is measured by 30-s chair-stand test
Upper limb strength | Assessments at baseline and at 6 weeks
  Upper limb strength is measured by hand grip strength tool
Quality of life | Assessments at baseline and at 6 weeks
  Quality of life is measured by World Health Organization Quality of Life HIV Instrument

IPD SHARING:
Plan to Share IPD: Undecided